CLINICAL TRIAL: NCT01798134
Title: Microparticle Enhanced Cytotoxic Transarterial Embolization Therapy in Hepatocellular Carcinoma
Acronym: MIRACLE I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TANDEM 2012-001 OUS
Record Dates: First submitted 2012-12-06; First posted 2013-02-25 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: To show safety; and efficacy; investigational product
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEB-TACE (Other): Transarterial Chemoembolization with TANDEM™ - DOX Microspheres (DEB-TACE)
  Treatment: Lobes; Dosing: TANDEM™/Doxorubicin; Second Treatment:TANDEM™/Doxorubicin
  Interventions: Device: TANDEM™

INTERVENTIONS:
Device: TANDEM™

SUMMARY:
This is a non-randomized, prospective, pilot, Multicenter Study of Drug-eluting bead transarterial chemoembolization (DEB-TACE) using Doxorubicin-Loaded Embozene® Tandem™ Microspheres to treat hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of HCC according to the European Association for the Study of the Liver (EASL) criteria for diagnosis, and staged according to the Barcelona clinic liver cancer (BCLC) criteria
2. Subject is competent and willing to provide written informed consent in order to participate in the study
3. Adults (male or female) patients ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or Child Pugh classification is 0-11
5. Multidonar or single nodular tumor ≥3-10cm, Patients with bilobar disease who can be treated superselectively in a single session or both lobes able to be treated within 3-5 weeks. Patient must have at least one tumor lesion that meets the following criteria: Lesion can be accurately measured in at least one dimension according to modified Response Evaluation Criteria In Solid Tumors (mRECIST) criteria
6. No invasion in the major blood vessel (hepatic portal, hepatic vein) or bile duct by the Magnetic resonance imaging (MRI) or Computed Tomography (CT)
7. Proper blood, liver, renal, heart function: testing result within 2 weeks from registry of this study
8. No current infections requiring antibiotic therapy
9. Not actively on cumarin based anticoagulation or suffering from a known bleeding disorder
10. Measurable disease per the Response Evaluation Criteria in Solid Tumors (mRECIST)
11. Expected survival more than 6 months

Exclusion Criteria:

1. ECOG performance status >2; or Child-Pugh class C11 or more, or ASA class 5
2. Bilirubin levels >3 mg/dl
3. HCC with large vessel or biliary duct invasion, diffuse HCC or extrahepatic spread
4. Patients in which any of the following are contraindicated or present:

   * The use of doxorubicin
   * MRI
   * Hepatic embolization procedures
   * White blood cell (WBC) < 3000 cells/mm3
   * neutrophil < 1500 cells/mm3
   * Cardiac ejection fraction < 50 percent assessed by isotopic ventriculography, echocardiography or MR
   * Elevated creatinine greater than or equal to 2.5 mg/dl
   * Impaired clotting test (platelet count < 5 x 104/mm3, Prothrombin time-International normalized ratio (PT-INR > 2.0)
   * aspartate transaminase (AST) and/or alanine transaminase (ALT) >5x ULN or, when greater >250 U/L
   * Known hepatofugal blood flow
   * Arterio-venous shunt
   * Arterio-portal shunt
   * Main stem portal vein occlusion(point 6 in inclusion criteria)
5. Women who are pregnant or breast feeding
6. Allergy to iodinated contrast used for angiography
7. Tumour burden of more than 50% of liver
8. Patients with objective signs of active bacterial, viral (human immunodeficiency virus (HIV)), or fungal infection
9. Other primary malignancies or evidence of metastatic disease
10. Patients previously treated with anthracyclines (other than doxorubicin).
11. Any co-morbid disease or condition or event that, in the investigator's judgment, would place the patient at undue risk that would preclude the safe use of DEB-TACE.
12. Under no circumstances should patients be enrolled in this study who is already participating in another study for treatment of primary liver cancer.
13. Under no circumstances should patients be enrolled in this study who has received any other embolotherapy (including Selective Internal Radiation Therapy (SIRT)) for the treatment of primary liver cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gotz M Richter, MD, Principal Investigator — Klinikum Stuttgart - Katharinenhospital
Locations (7):
- Germany (7):
  - Klinikum der Universitat Heidelberg, Heidelberg, Baden-Wurttemberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - Klinikum Stuttgart- Katharinenhospital, Stuttgart, Baden-Wurttemberg
  - Klinikum Bogenhausen, München, Bavaria
  - Kilinikum Darmstadt, Darmstadt, Hesse
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - University Hospital Regensburg, Regensburg

RESULTS

PARTICIPANT FLOW:
Groups:
- DEB-TACE: Transarterial Chemoembolization with TANDEM™ - DOX Microspheres (DEB-TACE)
  Treatment: Lobes; Dosing: TANDEM™/Doxorubicin; Second Treatment:TANDEM™/Doxorubicin
  TANDEM™
Period: Overall Study
Arm/Group | DEB-TACE
Started | 25
Completed | 9
Not Completed | 16
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 2
Not completed — Adverse Event | 3
Not completed — Physician Decision | 3
Not completed — Liver transplant/surgery | 4

BASELINE CHARACTERISTICS:
Arm/Group | DEB-TACE
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 65 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Serious Adverse Event (SAE) at 30days
Time Frame: Up to 30 days
Population: One participant is not included in the analysis as the investigator withdrew the participant 2 days after treatment started and then treated the participant systemically with sorafenib.
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 24
participants | 22

2. Primary Outcome: Freedom From Study Related SAE at 6 Months
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 24
participants | 21

3. Primary Outcome: Freedom From Tumor Progression at 6 Months
Description: Progression was assessed by the modified Response Evaluation Criteria in Solid Tumors (mRECIST - Lencioni and Llovet 2010) as an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: 6 months
Population: For efficacy outcomes, there were 21 participants with imaging to assess tumor response. No imaging was available for the other participants.
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 21
participants | 20

4. Secondary Outcome: 12 Month Survival
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 25
participants | 14

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DEB-TACE
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEB-TACE (N=25)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEB-TACE (N=25)
Abdominal pain (Gastrointestinal disorders) | 7 (12)
Abdominal pain upper (Gastrointestinal disorders) | 4 (8)
Angina pectoris (Cardiac disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood creatinine increased (Investigations) | 2 (3)
Blood potassium decreased (Investigations) | 2 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (7)
C-reactive protein increased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (10)
Oedema peripheral (General disorders) | 2 (3)
Pain (General disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pyrexia (General disorders) | 6 (8)
Urinary tract infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less